CLINICAL TRIAL: NCT04156906
Title: RH Genotype Matched Red Cells for Patients With Sickle Cell Disease and Anti-D
Brief Title: RHD Genotype Matched Red Cells for Anti-D
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: New York Blood Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-016566; R01HL147879-01 (NIH)
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease; Anti-D Antibodies
Keywords: Chronic Transfusion
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- D+ RH genotype matched Red Blood Cell Transfusion (Experimental): Investigators will provide one red cell unit of D+ RH genotype matched RBCs at the first transfusion study visit. The remainder of units will be provided per clinical standard of care, i.e. D-, CEK-matched, and negative for all other antigens the patient is alloimmunized against. If laboratory monitoring shows no reappearance of anti-D and no signs of increased red cell hemolysis, the patient will receive one unit of D+ RH genotype matched RBCs at the 2nd transfusion study visit, and if tolerated, D+ red cell exposures will increase by one unit per study visit until all units required are D+.
  Interventions: Biological: D+ RH genotype matched red cell units for transfusion

INTERVENTIONS:
Biological: D+ RH genotype matched red cell units for transfusion — Chronically transfused patients with SCD and anti-D will receive D+ RH genotyped matched red cell units for transfusion in addition to standard C, E, and K antigen matching and being hemoglobin S negative, which is the Children's Hospital of Philadelphia institutional standard of care for patients with SCD. RH genotyping of donor units will be performed by the New York Blood Center (NYBC) Immunogenetics laboratory.

SUMMARY:
This is a pilot study to evaluate the feasibility and safety of providing RH genotype matched D+ Red Blood Cells (RBCs) to chronically transfused patients with sickle cell disease (SCD) who type D+ but have formed anti-D and are currently transfused with D- RBC (Red Blood Cell) units.

DETAILED DESCRIPTION:
Red blood cell transfusion remains a critical therapy for patients with sickle cell disease (SCD). A major problem is the high rate of alloimmunization (antibody formation against transfused red cells) that occurs in patients with SCD. Recent studies performed by Investigators and others demonstrate RH genetic variants in patients and donors is a major risk factor leading to Rh alloimmunization. Anti-D formation in D+ patients occurs frequently, and once identified, providing D- cells for all subsequent transfusions can be challenging. These anti-D antibodies in D+ patients suggest exposure to different or variant D protein on donor cells. Investigators will test whether transfusion of patients with anti-D with RHD genotyped matched red cells is feasible, safe and can decrease D- donor unit demand.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age > 8 years old
* Diagnosis of SCD, all genotypes
* Require chronic red cell transfusion therapy
* History of anti-D
* RH genotype predicts D+ expression

Exclusion Criteria:

* Rare RH genotype that would preclude sufficient RBC units
* Antigen negative requirements due to alloimmunization that would preclude sufficient RBC units

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stella Chou, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Protected Health Information (PHI) will be shared with the New York Blood Center (NYBC) to order blood for the subjects. This will be done using a secure online blood ordering system. The NYBC uses an FDA-approved HIPAA secure system called Blood Enterprise Computer System (BECS) to store patient data and results, including PHI. 3rd party computers at New York Blood Center will also store study data using study identification (ID) numbers. The purpose of having study data coded at NYBC is for specialized testing for red antigens or antibodies for which we will provide some clinical data to assist in the laboratory evaluation. To assure that the transmission of data and samples maintains confidentiality we will used study ID numbers for these samples. The master list will be maintained at the Children's Hospital of Philadelphia (CHOP). The study databases are password protected and on password protected computers at CHOP and at NYBC, that are backed up on the research servers.
Supporting Information: Study Protocol
Time Frame: For the duration of the study
Access Criteria: Only study team members will have access to the data

REFERENCES:
- [Background] Chou ST, Jackson T, Vege S, Smith-Whitley K, Friedman DF, Westhoff CM. High prevalence of red blood cell alloimmunization in sickle cell disease despite transfusion from Rh-matched minority donors. Blood. 2013 Aug 8;122(6):1062-71. doi: 10.1182/blood-2013-03-490623. Epub 2013 May 30. PMID 23723452
- [Background] Vichinsky EP, Earles A, Johnson RA, Hoag MS, Williams A, Lubin B. Alloimmunization in sickle cell anemia and transfusion of racially unmatched blood. N Engl J Med. 1990 Jun 7;322(23):1617-21. doi: 10.1056/NEJM199006073222301. PMID 2342522
- [Background] Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014 Sep 10;312(10):1033-48. doi: 10.1001/jama.2014.10517. PMID 25203083
- [Background] Chou ST, Evans P, Vege S, Coleman SL, Friedman DF, Keller M, Westhoff CM. RH genotype matching for transfusion support in sickle cell disease. Blood. 2018 Sep 13;132(11):1198-1207. doi: 10.1182/blood-2018-05-851360. Epub 2018 Jul 19. PMID 30026182
- [Background] Dezan MR, Ribeiro IH, Oliveira VB, Vieira JB, Gomes FC, Franco LAM, Varuzza L, Ribeiro R, Chinoca KZ, Levi JE, Krieger JE, Pereira AC, Gualandro SFM, Rocha VG, Mendrone-Junior A, Sabino EC, Dinardo CL. RHD and RHCE genotyping by next-generation sequencing is an effective strategy to identify molecular variants within sickle cell disease patients. Blood Cells Mol Dis. 2017 Jun;65:8-15. doi: 10.1016/j.bcmd.2017.03.014. Epub 2017 Mar 31. PMID 28388467
- [Derived] Chou ST, Mewha J, Friedman DF, Lazariu V, Makrm S, Ochoa G, Vege S, Westhoff CM. Genotyped RhD+ red cells for D-positive patients with sickle cell disease with conventional RHD and unexpected anti-D. Blood. 2024 Nov 7;144(19):2045-2049. doi: 10.1182/blood.2024025602. PMID 39172743

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | D+ RH Genotype Matched Red Blood Cell Transfusion
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | D+ RH Genotype Matched Red Blood Cell Transfusion
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Anti-D Recurrence
Description: To determine safety of providing RH genotype match red cells to patients with a history of anti-D, we observed if anti-D reappearance occurred or evidence of hemolysis of transfused red cells.
Time Frame: Through study completion and follow-up phase, an average of 10 months per participant
Population: All participants completed all study requirements with no reappearance of anti-D.
Measure: Count of Participants; unit: Participants
Arm/Group | D+ RH Genotype Matched Red Blood Cell Transfusion
Number analyzed (Participants) | 5
Participants
  Anti-D recurrence | 0
  No anti-D recurrence | 5

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | D+ RH Genotype Matched Red Blood Cell Transfusion
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT04156906/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT04156906/ICF_001.pdf